CLINICAL TRIAL: NCT04824703
Title: Comparative Study Between Liberal and Conservative Oxygen Therapy in Mechanically Ventilated Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Sayed Mohamed Tammam, Assistant lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aswu/460/5/20
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Oxygen Therapy
Keywords: Oxygen therapy and Mortality
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conservative oxygen therapy (Active Comparator): * Spo2 alarm limit will be set as follow: - upper limit 94% and lower limit 88%
  * If spo2 >94% Unless fio2 is 0.21%, decrease fio2 by 0.10% at intervals no longer than 5 minutes till spo2 = 94%
  * If spo2 within target Decrease fio2 0.05% at intervals no longer than 30 min till fio2 0.21% reached or spo2 = 88 %
  * If spo2 < 88 % return to previous spo2 that achieve target spo2.
  * if an arterial blood gas demonstrate that the PaO2 is < 60 mmHg FiO2 will increased if clinically appropriate irrespective of the SpO2 reading ( target po2 60-100 mmhg )
  * During intubation, airway suction, tracheostomy, bronchoscopy, transportation outside of the ICU for radiological or other investigations or for procedures or operations, other critical situations such as hemodynamic collapse, patients will receive standard (non-study)treatment.
  * Echocardiography on randomization and at end of the study: we will calculate stroke volume according to Simpson's apical four view
  Interventions: Drug: Oxygen
- Liberal oxygen therapy (Placebo Comparator): * Spo2 target > 95%
  * No specific measures will be taken to avoid high fio2 or high po2
  * Use of upper alarm limit for spo2 will be prohibited
  * Echocardiography on randomization and at end of the study: we will calculate stroke volume according to Simpson's apical four view
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — * Decreasing fraction of inspired oxygen and its effect on mortality and myocardial function
  * administered by invasive mechanical ventilation with fraction of inspired oxygen between 0.21 and 1

SUMMARY:
To assess the benefits and drawbacks of high versus low oxygen therapy on mortality and myocardial function in mechanically ventilated patients

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years or older admitted to ICU and expected to receive mechanical ventilation beyond next calendar day

Exclusion Criteria:

* inclusion in other trial
* severe acute respiratory distress syndrome at time of admission
* acute Chronic obstructive airway disease exacerbation
* pregnancy
* Carbon monoxide poisoning
* Guillain Barre syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Change in Stroke volume in milliliters | Change from Baseline stroke volume At ICU admission and through study completion An average 6 months
  Volume of blood in milliliters that is ejected from heart each second and measured By Echocardiography
Change in ejection fraction of heart in percentage | Change from baseline ejection fraction at icu admission and through study completion An Average 6 months
  percentage of blood that's pumped out of a filled ventricle with each heartbeat And measured by echocardiography

SECONDARY OUTCOMES:
Acute respiratory distress syndrome | From icu admission date to icu discharge date an average of 2 weeks
  Acute persistent hypoxia with bilateral lung infiltrate due to non cardiac cause
Sepsis | From icu admission date to icu discharge date an average of 2 weeks
  Systolic blood pressure < 90 Respiratory rate > 22 Heart rate > 100
Stroke | From icu admission date to icu discharge date an average of 2 weeks
  Cerebrovascular accidents
Mechanical Ventilator free days | From icu admission date to icu discharge date an average of 2 weeks
  Days without mechanical ventilation
Shock | From icu admission date to icu discharge date an average of 2 weeks
  Systolic blood pressure < 90 mmHg
Surgery revision | From icu admission date to icu discharge date an average of 2 weeks
  Surgical re exploration
Vasopressor | From icu admission date to icu discharge date an average of 2 weeks
  Use of vasopressors as norepinephrine and epinephrine
ICU stay | From icu admission date to icu discharge date an average of 2 weeks
  Duration of intensive care stay
Hospital stay | From icu admission date to icu discharge date an average of 2 weeks
  Duration of hospital stay
Mortality | From icu admission date to icu discharge date an average of 2 weeks
  Death of patient

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan university hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ghazaly HF, Aly AAA, Tammam AS, Hassan MM, Hammad SS, Mahmoud NM, Hemaida TS. Influence of liberal versus conservative oxygen therapies on the hemodynamic parameters of mechanically ventilated patients with sepsis: a randomized clinical trial. BMC Anesthesiol. 2024 Dec 20;24(1):469. doi: 10.1186/s12871-024-02838-6. PMID 39707209